CLINICAL TRIAL: NCT05904938
Title: Efficacy and Safety of Oral Administration of the Plant-based Complex Actitan-F in the Management of Chronic Paediatric Diarrhoea: a Double-blind, Placebo-controlled, Parallel-group Investigation
Brief Title: Oral Administration of Actitan-F in Paediatric Diarrhoea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: IQVIA RDS Inc. (Industry); IQVIA Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABO-LENP-01/22
Record Dates: First submitted 2023-03-16; First posted 2023-06-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-06

CONDITIONS: Chronic Diarrhoea of Infants and/or Young Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenodiar Pediatric (Experimental): Medical Device
  Interventions: Device: Lenodiar Pediatric
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Lenodiar Pediatric — Medical Device made of natural substance
  Arms: Lenodiar Pediatric
Other: Placebo — Product appearance similar to verum without clinical efficacy
  Arms: Placebo

SUMMARY:
The goal of the study is to investigate the efficacy and safety of Lenodiar Pediatric (product under investigation) for the treatment of Chronic Diarrhoea (functional or post-infective diarrhoea) in children aged 1-5 years old, through a randomized, double blind, placebo-controlled clinical investigation

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged between 1-5 years (inclusive);
* Diagnosis of chronic diarrhoea due to the following conditions:

  * Functional gastrointestinal disorder fulfilling Rome IV Criteria*
  * or
  * Functional gastrointestinal disorder fulfilling modified Rome IV Criteria **
  * or
  * Post-infectious diarrea with daily painless, recurrent passage of three or more large, unformed stools
* Parents/legal guardians*** availability to fill on a daily basis the electronic daily diary by a smartphone/tablet.
* Parents/legal guardians have given a written informed consent for participation in the investigation at the time of enrolment or before. The parent/legal guardian should also have agreed to bring the child for the visits scheduled in the protocol and to provide the requested information during the telephonic follow-up visit;
* Parents/legal guardian able to understand the full nature and the purpose of the investigation, including possible risks and side effects, able to cooperate with the Investigator and to comply with the requirements of the entire investigation (ability to attend all the planned investigation visits according to the time limits included) based on Investigator's judgement;
* Willingness not to make diet and lifestyle significant changes during the trial.

  * Rome IV criteria of functional diarrhoea (Neonate and Toddlers below 5 years), must include all of the following:

    * Daily painless, recurrent passage of four or more large, unformed stools
    * Symptoms last more than 4 weeks
    * Onset between 6 and 60 months of age
    * No failure-to-thrive if caloric intake is adequate

      ** Modified Rome IV criteria of functional diarrhoea (Neonate and Toddlers below 5 years), must include all of the following:
    * Daily painless, recurrent passage of three or more large, unformed stools
    * Symptoms last more than 2 weeks (Nelson Pediatric Texbook 21st Edition, Chronic diarrhea)
    * Onset between 6 and 60 months of age
    * No failure-to-thrive if caloric intake is adequate
    * These criteria have been modified in order to align the study to the functional diarrhoea condition in the real life.

      * Parent is the child's biological or adoptive parent. Legal guardian is defined as an individual who was authorized under applicable state or local law to consent on behalf of a child to general medical care, when general medical care includes participation in research. A guardian also meant an individual who was authorized to consent on behalf of a child to participate in research.

Exclusion Criteria:

* Carbohydrate malabsorption, diagnosed either clinically (2 weeks exclusion diet with resolution of symptoms) or with proper testing (breath test)*;
* Patients with any of the following chronic gastrointestinal disorders: inflammatory bowel disease, pancreatitis, chronic liver disease, eosinophilic oesophagitis, peptic ulcer disease, celiac disease, pseudo-obstruction, small bowel bacterial overgrowth, or Hirschsprung's disease
* Significant chronic health condition requiring specialty care (e.g., lithiasis, ureteropelvic junction obstruction, sickle cell, cerebral palsy, hepatic, hematopoietic, renal, endocrine, or metabolic diseases) that could potentially impact the child's ability to participate or confound the results of the investigation;
* Gastrointestinal blood loss;
* Recurrent or unexplained fevers;
* Developmental disabilities impairing ability to understand or communicate;
* History of hypersensitivity or allergy to investigational product;
* History of previous abdominal surgeries in the past 3 months;
* Known hypersensitivity to any of the components (active ingredients or excipients) of the investigational product;
* Conditions known to producing immunodeficiency (AIDS, other congenital immunodeficiency syndromes, drugs therapy with steroids, anticancer drugs, etc.);
* Patients who have received any of the following treatments within the 2 weeks before the baseline visit:

  * Agents specially developed for achieving adsorbing properties, e.g. kaolin, pectin, bismuth subsalicylate;
  * Treatments that modify intestinal secretions, e.g. racecadotril;
  * Treatments that modify intestinal motility, e.g. opiates, anti-cholinergic agents;
  * Systemic Antibiotics;
  * Antiemetic agents.
* Patients who have received probiotics and prebiotics within the 1 week before the baseline visit, unless they have been taken at stable dose (the use of probiotics and prebiotics in dairy food such as yoghurt, cheese, milk prior to the investigation is permitted);
* Parents/legal guardians' refusal or inability to give written informed consent to participate in the investigation;
* Parents/legal guardians who, in the opinion of the Investigator, are unable to fill up the electronic patient diary;
* Patients who have participated in any other clinical trial in the last 3 months prior to the start of the investigation.

  * Applicable only for patients with Functional gastrointestinal disorder fulfilling Rome IV Criteria.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in stool consistency averaged over the 2-week Treatment Period | Up to 2 weeks vs Baseline
  Stool consistency will be assessed using the Bristol Stool Form Scale (BSFS) on a range from 1 (Hard Lumps) to 7 (Watery).

SECONDARY OUTCOMES:
Change for daily daytime and nighttime stool consistency scores | (Week1 to Week4) vs Baseline
  Change for daily daytime and nighttime stool consistency scores assessed using the Bristol Stool Form Scale (BSFS) on a range from 1 (Hard Lumps) to 7 (Watery).
Change for 24-hour abdominal pain scores | (Week1 to Week4) vs Baseline
  Abdominal Pain is scored on a five-point ordinal scale, with 0 meaning no pain, and 4 meaning a lot of pain.
Change for daytime, nighttime, and 24-hour bowel movement frequency | (Week1 to Week4) vs Baseline
  Change for daytime, nighttime, and 24-hour bowel movement frequency
Change for daytime, nighttime, and 24-hour urgency-free days | (Week1 to Week4) vs Baseline
  Change for daytime, nighttime, and 24-hour urgency-free days (only for patients who have removed the diaper and have received training toilet)
Time to event, with the event defined as the first week in which a reduction ≥50% of loose or watery stools as compared to baseline occurs. | through study completion, an average of 4 weeks
  Time to event is defined as the time elapsed (days) from the date of randomization to the date of the first week in which a reduction ≥50% of loose or watery stools as compared to baseline occurs. This endpoint will be assessed through electronic diary.
Use of other treatments (proportion of users) for diarrhea relief, evaluated by means of the electronic patient diaries; | through study completion, an average of 4 weeks
  Use of other treatments (proportion of users and quantity) for diarrhea relief, evaluated through a electronic patient diaries;
Use of other treatments (quantity of other treatments) for diarrhea relief, evaluated by means of the electronic patient diaries; | through study completion, an average of 4 weeks
  Use of other treatments (proportion of users and quantity) for diarrhea relief, evaluated through a electronic patient diaries;
Change in results of the Pediatric Quality of Life Questionnaires | Visit 1 (day 14); Visit 2 (day 28);
  Change in results of the Pediatric Quality of Life Questionnaires assessed through a validated questionnaire
Change in results of the patient happiness using a weekly smiley likert scale | through study completion, an average of 4 weeks
  Parents/legal guardians will report, on a weekly basis, the happiness of the patients using a smiley face likert scale (Very happy; Happy; Slightly happy; Neutral; Slightly unhappy)
Change in results in parent Quality of Life (100 mm VAS) | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change in results in parent Quality of Life using a 100 mm Visual Analogie Scale, ranging from "0" (corresponds to a quality of life "very low") and the value "100" (corresponds to a quality of life "very high")
Time to event, with the event defined as the first day in which loose or watery stools are not observed. | through study completion, an average of 4 weeks
  Time to event is defined as the time elapsed (days) from the date of randomization to the date of the first day in which loose or watery stools are not observed.
Change in patients' lifestyle | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change in patients' lifestyle assessed through a lifestyle questionnaire
Time to event, with the event defined as the third day of the first consecutive three days in which diagnostic criteria for chronic diarrhoea are no more met. | through study completion, an average of 4 weeks
  Time to event is defined as the time elapsed (days) from the date of randomization to the date of the third of the first consecutive three days in which diagnostic criteria for chronic diarrhoea are no more met
Change from baseline in stool consistency at day 3, day 7 and day 10. | Baseline to day 3, day 7 and day 10
  Change from baseline in stool consistency at day 3, day 7 and day 10. Stool consistency will be assessed using the Bristol Stool Form Scale (BSFS) on a range from 1 (Hard Lumps) to 7 (Watery).
Adverse Event | through study completion, an average of 4 weeks
  Incidence of adverse events (AEs)
Serious Adverse Event | through study completion, an average of 4 weeks
  Incidence of serious adverse events (SAEs)
Adverse device effects | through study completion, an average of 4 weeks
  Incidence of adverse device effects (ADEs)
Serious adverse device effects | through study completion, an average of 4 weeks
  Incidence of a serious adverse device effects (SADEs)
Unexpected serious adverse device effects | through study completion, an average of 4 weeks
  Incidence of unexpected serious adverse device effects (USADEs)
Early withdrawal rate due to AEs | through study completion, an average of 4 weeks
  Incidence of early withdrawal rate due to AEs, whether serious or not
Safety Endpoints - early withdrawal rate due to ADEs | through study completion, an average of 4 weeks
  Incidence of early withdrawal rate due to ADEs, whether serious or not.
Systolic/diastolic blood pressure | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change from baseline in clinical examination findings (systolic/diastolic blood pressure)
Pulse | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change from baseline in clinical examination findings (pulse)
Weight | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change from baseline in clinical examination findings (weight)
Body Mass Index | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change from baseline in clinical examination findings (Body Mass Index)
Waist circumference | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Change from baseline in clinical examination findings (waist circumference)

OTHER OUTCOMES:
Faecal microbiota | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Differences before and after treatment in the analyses of Faecal microbiota, collecting and analysing stool samples
Faecal metabolomics | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Differences before and after treatment in the analyses of Faecal metabolomics, , collecting and analysing stool samples.
Micro RNA | Baseline to Visit 1 (day 14) and Visit 2 (day 28) and Visit 1 (day 14) to Visit 2 (day 28)
  Differences before and after treatment in the analyses of Micro RNA (miRNA) from mouth epithelial cells, , collecting and analysing buccal samples

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Azienda Ospedaliera Universitaria "Federico II",, Napoli, Italia
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Cannizzaro, UOC Pediatria e PS Pediatrico, Catania
  - Policlinico "SS. Annunziata" Clinica Pediatrica Via dei Vestini, Località colle dell'Ara 66100, Chieti, Chieti
  - IRCCS AOU Meyer SOC Gastroenterologia e Nutrizione, Viale Gaetano Pieraccini 24, Florence
  - Azienda Socio Sanitaria Territoriale Santi Paolo e Carlo Presidio San Carlo, Ambulatorio di Gastroenterologia Pediatrica, Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", I Clinica Pediatrica, Napoli
  - ARNAS Ospedale Civico e Benfratelli G Cristina e M Ascoli, Pediatria ad Indirizzo Gastroenterologico, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pediatria, Pavia
  - Ospedale S. Maria della Misericordia, Perugia
  - Ospedale San Jacopo di Pistoia, SOC Pediatria, Pistoia
  - U.O. di Gastroenterologia e Riabilitazione Nutrizionale Ospedale Pediatrico Bambin Gesu Piazza S. Onofrio, 4 00165, Roma, Roma